CLINICAL TRIAL: NCT00870571
Title: Comparative, Randomized, Single Dose, 2-way Crossover Bioavailability Study of Actavis Group hf and Pfizer Inc. (Norvasc®)10 mg Amlodipine Besylate Tablets in Healthy Adult Volunteers Under Fed Conditions.
Brief Title: A Relative Bioavailability Study of Amlodipine Besylate 10 mg Tablets Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 24309
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; amlodipine besylate; amlodipine; Healthy subjects
MeSH Terms: interventions — Amlodipine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AMLODIPINE (as BESILATE) TABLETS 10 mg, single dose
  Interventions: Drug: AMLODIPINE (as BESILATE) TABLETS 10 mg , single dose
- B (Active Comparator): NorvasC® 10 mg Tablets, single dose
  Interventions: Drug: NorvasC® 10 mg Tablets

INTERVENTIONS:
Drug: AMLODIPINE (as BESILATE) TABLETS 10 mg , single dose — A: Experimental Subjects received EMCURE PHARMACEUTICALS LTD. formulated products under fed conditions
  Other Names: amlodipine besylate; amlodipine
  Arms: A
Drug: NorvasC® 10 mg Tablets — B: Active comparator Subjects received Pfizer Labs Division of Pfizer Inc. formulated products under fed conditions
  Other Names: amlodipine besylate; amlodipine
  Arms: B

SUMMARY:
The purpose of this study to assess the single-dose relative bioavailability of Actavis Group hf and Pfizer (Norvasc®) 10 mg amlodipine besylate tablets, under fed conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Actavis Group hf and Pfizer Inc. (Norvasc®) 10 mg Amlodipine Besylate Tablets in Healthy Adult Volunteers under FedConditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

Subject candidates must fulfill all of the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

* Healthy adult male or female volunteers, 18-55 years of age;
* Subject will be non-smokers or moderate smokers (less than 10 cigarettes a day) for at least 3 months.
* Weighing at least 60 kg for males and 52 kg for females and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983);
* Medically healthy subjects with clinically normal laboratory profiles. vital signs and ECGs;
* Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the first dose, throughout the study and for 14 days following the last dose or be using one of the following acceptable birth control methods:

  1. surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum.
  2. IUD in place for at least 3 months.
  3. barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose, throughout the study, and for 14 days following the last dose.
  4. surgical sterilization of the partner (vasectomy for 6 months minimum).
  5. hormonal contraceptives for at least 3 months prior to the first dose of the study and for 14 days following the last dose.

     Other birth control methods may be deemed acceptable. Postmenopausal women with amenorrhea for at least 2 years will be eligible.
* Give voluntary written informed consent to participate in the study.

Exclusion Criteria:

* Subject candidates must not be enrolled in the study if they meet any of the following criteria:
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of:
* alcoholism or drug abuse within the past year;
* hypersensitivity or idiosyncratic reaction to amlodipine or other calcium channel blockers.
* Female subjects who are pregnant or lactating.
* SUbjects who tested positive at screening for HIV, HbsAg or HeV.
* Subjects whose sitting blood pressure is less than 110/60 mmHg at screening or 100/55 mmHg before dosing.
* Subjects whose pulse is lower than 55 b.p.m. at screening or 50 b.p.m. prior to dosing.
* Subjects who have used any drugs or substances known to be strong inhibitors of CYP enzymes (formerly known as cytochrome P450 enzymes) within 10 days prior to the first dose.
* Subjects who have used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
* Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who, through completion of the study, would have donated in excess of: 500 mL of blood In 14 days; 1500 mL of blood in 160 days; 2500 mL of blood In 1 year.
* Subjects who have participated in another clinical trial within 28 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2005-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli,, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Saint-Laurent, Montreal, Quebec, Canada